CLINICAL TRIAL: NCT01350011
Title: Extended Tobacco Dependence Intervention in Buprenorphine Treatment
Brief Title: Tobacco Intervention in Buprenorphine Treatment
Acronym: IBIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P030871; P50DA009253 (NIH)
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Tobacco Dependence
Keywords: Nicotine Replacement Therapy; Buprenorphine; Varenicline; Smoking Cessation; Addiction; The Innovative System (IS) Treatment; The Standard Treatment Control (STC)
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Innovative System (IS) (Active Comparator): The innovative intervention uses the treatment system to support motivational counseling treatment entrance and treatment utilization. It has two components, a Motivational Intervention component via Expert System Counseling, and a Treatment Component that incorporates both pharmacological and behavioral long-term components. An innovative aspect of the IS is the use of the pharmacist as an intervention agent, who queries participants on their readiness to quit smoking, encourages involvement in the motivational intervention and in treatment, and who, along with the counselors, is available to answer medication questions.
  Interventions: Behavioral: Innovative System
- Standard Treatment Control (Active Comparator): After a baseline interview, patients in this condition will be given a packet of brochures on quitting, including descriptions of self-quitting and help-lines. Participants in this condition will continue to have access to their primary care providers, and through that system have access to pharmacotherapy for smoking cessation, if they wish to receive it. They will receive written instructions on how to approach their primary care provider about smoking cessation medication, and a written description of the medications used in smoking cessation and a list of those that are available to them through the public health system. At each assessment, patients will be queried about their use of these resources.
  Interventions: Behavioral: Standard Treatment Control (STC)

INTERVENTIONS:
Behavioral: Innovative System — In IS, they will receive motivational counseling at months 3,6,12, and 18. If they decide to quit smoking they will be offered up to 10 sessions of behavioral counseling and access to NRT (nicotine patch and gum) If they relapse on NRT, they will be offered varenicline, if it is not contraindicated.
  Arms: Innovative System (IS)
Behavioral: Standard Treatment Control (STC) — Participants will receive self help information and referrals for counseling and for pharmacological treatment.
  Arms: Standard Treatment Control

SUMMARY:
Drug addiction treatment patients, including those in treatment for opioid dependence, have a high rate of tobacco dependence, especially cigarette smoking. The proposed study evaluates an Innovative System (IS) for the treatment of tobacco dependence in one group of opioid treatment patients, those in buprenorphine maintenance. The specific aims of the study are to test the efficacy and the cost effectiveness of the IS.

A secondary aim is obtain preliminary data about differences in use of non-nicotinic drugs between participants who achieve abstinence from cigarettes during the study, and those who do not.

DETAILED DESCRIPTION:
This component is grounded in the past work of the Center. It continues the tradition of working with complex populations in new settings. However, it addresses the problem that shorter (standard or traditional tobacco dependence) interventions do not appear to work well in this population, and it tests a research-based alternative that has shown effectiveness in prior research. If the Innovative System (IS) that we propose is shown to be effective in this population, this line of research will offer the field a strategy to more effectively address tobacco dependence among persons with non-nicotinic drug abuse disorders. It is an extended treatment, and with appropriate adaptations, could become a continuing care intervention in a variety of health systems using a variety of health care personnel, including pharmacists, primary care physicians & nurses.

Drug addiction treatment patients, including those in treatment for opioid dependence, have a high rate of tobacco dependence, especially cigarette smoking. The proposed study evaluates an Innovative System (IS) for the treatment of tobacco dependence in one group of opioid treatment patients, those in buprenorphine maintenance. The primary specific aims of the proposed study are to test four efficacy hypotheses and to study cost and cost effectiveness of the IS. We will test the following four hypotheses and explore one additional primary aim:

1. We hypothesize that at months 12 and 18, participants in IS will attain higher biochemically verified cigarette abstinence rates than those in STC.
2. We hypothesize that at months 6, 12, and 18, participants in IS will report more quit attempts and more stringent cigarette abstinence goals than participants in STC.
3. We hypothesize that, in both treatment conditions, a higher number of cigarettes smoked at baseline and higher baseline Fagerström Test of Nicotine Dependence (FTND) score will predict a lower probability of abstinence at months 3, 6, 12, and 18.
4. We hypothesize that, in both experimental conditions, participants with smaller Cotinine/3HC (COT/3HC) ratios will be more likely to be abstinent at months 3, 6, 12, and 18, than those with larger ratios.
5. The final primary specific aim is to determine the cost of providing innovative smoking cessation treatment to opiate dependent individuals in buprenorphine treatment and to learn if the treatment is cost-effective, that is, if its benefits are sufficient to justify its cost. This aim reflects an ongoing and historical emphasis in this P50 center grant, that of obtaining cost and cost-effectiveness data, as well as efficacy data A secondary aim is to obtain preliminary data about differences in use of non-nicotinic drugs between participants who achieve abstinence from cigarettes during the study, and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* All participants must smoke five or more cigarettes a day and be registered patients at Integrated Buprenorphine Intervention Services (IBIS) of the San Francisco Department of Public Health.

Exclusion Criteria:

* Participants with contraindications to NRT will be excluded. Thus, participants who have had a myocardial infarction within the last three months, or who have uncontrolled high blood pressure will be excluded. We will exclude pregnant or nursing women.
* Participants with contraindications to varenicline treatment will be included in the study but will not be eligible for varenicline treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Smoking Status | 3, 6, 12, and 18 Months
  Smoking status is defined as "no cigarettes for the past 7 days."

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hall, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Behavioral Health Access Center, San Francisco, California, United States

REFERENCES:
- [Derived] Hall SM, Humfleet GL, Gasper JJ, Delucchi KL, Hersh DF, Guydish JR. Cigarette Smoking Cessation Intervention for Buprenorphine Treatment Patients. Nicotine Tob Res. 2018 Apr 2;20(5):628-635. doi: 10.1093/ntr/ntx113. PMID 28549161